CLINICAL TRIAL: NCT00277160
Title: A Randomized, Open Label, Multicenter Study of Primary Prophylaxis With Neulasta (Pegfilgrastim) Versus Secondary Prophylaxis as an Adjunct to Chemotherapy in Elderly Subjects (>/= 65 Years Old) With Cancer
Brief Title: A Study of Primary Prophylaxis With Neulasta (Pegfilgrastim) Versus Secondary Prophylaxis After Chemotherapy in Elderly Subjects (>/= 65 Years Old) With Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20020122
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2010-10-08 (Estimated); Status verified 2010-10

CONDITIONS: Neutropenia; Breast Cancer; Lung Cancer; Non-Hodgkin's Lymphoma; Ovarian Cancer
MeSH Terms: conditions — Neutropenia; Breast Neoplasms; Lung Neoplasms; Lymphoma, Non-Hodgkin; Ovarian Neoplasms | interventions — pegfilgrastim

ARMS (2):
- Treatment Group 1 (Primary Prophylaxis) (Experimental): Neulasta 6mg single administration per cycle of chemotherapy starting with cycle 1
  Interventions: Drug: Neulasta (pegfilgrastim)
- Treatment Group 2 (Secondary Prophylaxis) (Active Comparator): Per Investigator's discretion
  Interventions: Drug: Neulasta (pegfilgrastim)

INTERVENTIONS:
Drug: Neulasta (pegfilgrastim) — Commercial pegfilgrastim 6mg single subcutaneous fixed-dose

SUMMARY:
The purpose of this study is to assess pegfilgrastim starting with the first cycle versus secondary prophylaxis on neutropenic events (including neutropenia +/- fever, dose delays, dose reductions, and hospitalizations) in older patients receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* >/= 65 years old
* documented diagnosis of lung, breast, or ovarian cancer, or NHL
* scheduled to receive one of 15 standard chemotherapy regimens
* chemotherapy naive OR have received adjuvant therapy AND/OR have no more than one regimen of chemotherapy for metastatic disease
* life expectancy of at least 3 months
* ECOG performance status </=2
* adequate renal and hematologic function
* informed consent for participation in the study prior to any study specific procedures

Exclusion Criteria:

* known hypersensitivity to any of the products to be administered during dosing
* primary prophylactic antibiotics in all cycles
* prior radiation therapy within 2 weeks of randomization into this study or plan for radiation therapy during study participation, except for spot radiation for bony metastases
* prior bone marrow or stem cell transplant or plan to receive any transplant therapy during study participation
* clinically symptomatic brain metastases
* Folstein mini-mental state exam score <18
* Any premalignant myeloid condition or any malignancy with myeloid characteristics
* History of prior malignancy within the last 5 years other than subject's original cancer diagnosis listed in inclusion criteria with the exception of curatively treated basal cell carcinoma, squamous cell carcinoma, in situ cervical carcinoma or surgically cured malignancies
* unstable/uncontrolled cardiac conditions or hypertension
* active infection
* subject is currently enrolled or has not yet completed at least 30 days since ending other investigational device or drug trial or is receiving other investigational agents

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 852 (Actual)
Dates: Start 2002-06; Primary Completion 2004-11 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Incidence of febrile neutropenia, defined by ANC < 1.0 x 10^9/L and temperature ≥ 38o C on the same day | End of the last cycle of chemotherapy or the date of early termination from the study

SECONDARY OUTCOMES:
Incidence of grade 3 and 4 neutropenia | End of the last cycle of chemotherapy or the date of early termination from the study
Dose delays or dose reductions | End of the last cycle of chemotherapy or the date of early termination from the study
Incidence of febrile neutropenia with a more strict definition (ANC < 0.5 x 10^9/L and temperature ≥ 38o C), on the same day | End of the last cycle of chemotherapy or the date of early termination from the study

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Balducci L, Al-Halawani H, Charu V, Tam J, Shahin S, Dreiling L, Ershler WB. Elderly cancer patients receiving chemotherapy benefit from first-cycle pegfilgrastim. Oncologist. 2007 Dec;12(12):1416-24. doi: 10.1634/theoncologist.12-12-1416. PMID 18165618
- [Result] Flores IQ, Ershler W. Managing neutropenia in older patients with cancer receiving chemotherapy in a community setting. Clin J Oncol Nurs. 2010 Feb;14(1):81-6. doi: 10.1188/10.CJON.81-86. PMID 20118030
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com